CLINICAL TRIAL: NCT05224609
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL-GROUP STUDY TO EVALUATE THE PLASMA PHARMACOKINETICS AND SAFETY OF LORLATINIB IN PARTICIPANTS WITH MODERATE AND SEVERE HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
Brief Title: A Study to Learn About the Study Medicine (Called Lorlatinib) in People With Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B7461040
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Moderate Hepatic Impairment; Severe Hepatic Impairment; Healthy Volunteers
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Moderate hepatic impairment group
  Interventions: Drug: Lorlatinib
- Cohort 2 (Experimental): Severe hepatic impairment group
  Interventions: Drug: Lorlatinib
- Cohort 3 (Experimental): Normal hepatic function
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Single 100mg oral dose anti-cancer agent
  Other Names: Lorbrena; PF-06463922

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called Lorlatinib) in health participants. This study is seeking participants who:

* Must be male or female of 18 to 75 years of age, inclusive at the time of the study.
* Are willing and able to comply with all scheduled visits, treatment plan, and other study procedures.
* Have a BMI (body mass index) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb).
* Are capable of giving signed informed consent document. All participants in this study will receive Lorlatinib. Participants will be placed into 1 of 3 cohorts based on their hepatic (liver) function. Participants will take Lorlatinib once by mouth. We will examine the experiences of people receiving the study medicine. This will help us determine if the study medicine is safe and effective. Participants will take part in this study for up to 35 days.

DETAILED DESCRIPTION:
This is a Phase 1, open label, parallel group study to investigate the effect of moderate and severe hepatic impairment on the plasma PK, safety, and tolerability after a single oral 100 mg dose of lorlatinib under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

All Participants -

1. Participants must be male or female of 18 to 75 years of age, inclusive, at the time of signing the ICD.
2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. BMI of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb).
4. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Additional Inclusion Criteria for Participants with Normal Hepatic Function (Cohort 3) -

1. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, including BP and pulse rate measurement, 12-lead ECG or clinical laboratory tests. Particularly, should confirm no known or suspected hepatic impairment based on liver function tests (eg, ALT, AST, ALP, and bilirubin), albumin and prothrombin time.
2. Participants must fit the demographic-matching criteria, including: Body weight +- 15 kg of the median of the combined moderate and severe hepatic impairment cohorts (Cohorts 1 and 2), as provided by the sponsor.

Age +- 10 years of the median of the combined moderate and severe hepatic impairment cohorts (Cohorts 1 and 2), as provided by the sponsor.

Comparable male/female ratio to moderate and severe hepatic impairment cohorts (Cohorts 1 and 2).

Additional Inclusion Criteria for Participants with Moderately Impaired Hepatic Function (Cohort 1) -

1. Meet the criteria for Class B (moderate hepatic impairment) of the modified Child-Pugh classification.
2. A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography scan, or MRI.
3. Stable hepatic impairment, defined as no clinically significant known change in disease status within the last 30 days, as documented by the participant's recent medical history (eg, no worsening clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time by more than 50%).
4. Stable drug regimen is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to the dosing of lorlatinib.
5. History of alcohol abuse is permissible providing that the results of alcohol test are negative at Screening or on Day -1, and the participant is willing and able to abide by the lifestyle guidelines.

Additional Inclusion Criteria for Participants with Severely Impaired Hepatic Function (Cohort 2) -

1. Meet the criteria for Class C (severe hepatic impairment) of the modified Child-Pugh classification.
2. A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography scan, or MRI.
3. Stable hepatic impairment, defined as no clinically significant known change in disease status within the last 30 days, as documented by the participant's recent medical history (eg, no worsening clinical signs of hepatic impairment, or no worsening of TBili or prothrombin time by more than 50%).
4. Stable drug regimen is defined as not starting a new drug or changing dosage within 7 days or 5 half lives (whichever is longer) prior to the dosing of lorlatinib.
5. History of alcohol abuse is permissible providing that the results of alcohol test are negative on Screening or on Day -1, and the participant is willing and able to abide by the lifestyle guidelines.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

All Participants -

1. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
2. History of or current positive results for HIV infection.
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg. Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. Participants with an eGFR of ≤ 60 mL/min/1.73 m2 based on the 2021 CKD-EPI equation, with a single repeat permitted to assess eligibility, if needed.
5. Concurrent use of any of the following prohibited concomitant medication(s) within 12 days prior to the first dose of lorlatinib:

   1. Known strong CYP3A inhibitors (eg, boceprevir, cobicistat, clarithromycin, conivaptan, diltiazem, idelalisib, indinavir, itraconazole, ketoconazole, lopinavir, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, tipranavir, troleandomycin, voriconazole, grapefruit juice or grapefruit/grapefruit-related citrus fruits [eg Seville oranges, pomelos]). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
   2. Known strong CYP3A inducers (eg, carbamazepine, enzalutamide, mitotane, phenytoin, rifabutin, rifampin, St. John's Wort).
   3. Known P-gp substrates with a narrow therapeutic index (eg, digoxin).
6. Concurrent use of CYP3A substrates with narrow therapeutic indices (eg, alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl including transdermal patch, pimozide, quinidine, sirolimus, tacrolimus) within 12 days prior to the first dose of lorlatinib.
7. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
8. Known hypersensitivity to lorlatinib or its excipients.
9. A positive urine drug test. Participants with moderate or severe hepatic impairment (Cohorts 1 and 2) will be eligible to participate if their urine drug test is positive with a drug for a prescribed condition that is not expected to interfere with the PK of lorlatinib.
10. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
11. History of sensitivity to heparin or heparin-induced thrombocytopenia.
12. Unwilling or unable to comply with the criteria in the Lifestyle Considerations,
13. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Additional Exclusion Criteria for Participants with Normal Hepatic Function (Cohort 3) -

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies deemed relevant for participation in this study, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
3. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If initial supine BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
4. Baseline standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, baseline PR interval >200, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
5. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of nonprescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case by case basis following approval by the Sponsor. Herbal supplements and HRT must have been discontinued at least 28 days prior to the dose of lorlatinib.
6. Participants with a history of or current positive results for hepatitis B or hepatitis C, including HBsAg, HBcAb, or HCVAb.

Additional Exclusion Criteria for Participants with Moderate and Severe Hepatic Impairment (Cohorts 1 and 2) -

1. Other clinically significant disease that contraindicates study drug or that may affect the PK of lorlatinib.
2. Hepatic carcinoma and hepatorenal syndrome.
3. Undergone porta-caval shunt surgery.
4. History of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 1 month prior to study entry.
5. Any clinically significant laboratory abnormality except for those parameters influenced by hepatic impairment.
6. Presence of clinically active Stage 2, 3 or 4 encephalopathy.
7. Severe uncontrolled ascites and/or pleural effusion.
8. Screening supine BP ≥160 mm Hg (systolic) or ≥90 mm Hg (diastolic), on a single measurement following at least 5 minutes of rest. If initial supine BP is ≥160 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the three BP values should be used to determine the participant's eligibility.
9. Screening supine 12-lead ECG demonstrating QTcF >470 msec. If initial QTcF exceeds 470 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the participant's eligibility.
10. Second-degree or third-degree AV block (unless paced) or baseline PR interval >200 msec at any time prior to dosing of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Single dose Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (inf)] of lorlatinib | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post-dose
  PK parameter of lorlatinib to be calculated from the plasma concentration time data.
Single dose Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (last)] of lorlatinib | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post-dose
  PK parameter of lorlatinib to be calculated from the plasma concentration time data.
Single dose Maximum Observed Plasma Concentration (Cmax) of lorlatinib | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post-dose
  Maximum lorlatinib plasma concentration observed during study.

SECONDARY OUTCOMES:
Number of participants experienced treatment emergent adverse event assessed by investigator | Baseline up to Day 35
  Type, incidence, severity, seriousness, and relationship to study medications of adverse events (AE)
Number of participants experienced treatment related adverse event assessed by investigator | Baseline up to Day 35
  Type, incidence, severity, seriousness, and relationship to study medications of adverse events (AE)
Number of participants experienced serious adverse event assessed by investigator | Baseline up to Day 35
  Type, incidence, severity, seriousness, and relationship to study medications of adverse events (AE)
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Day 35
  Vital signs (pulse, systolic and diastolic blood pressure) were obtained. Clinical significance of vital signs was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Day 8
  Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell count, MCV, MCH, MCHC, platelet count, white blood cell count, neutrophils, eosinophils, monocytes, basophils, and lymphocytes), chemistry (blood urea nitrogen, creatinine, glucose [fasting], calcium, sodium, potassium, chloride, bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, direct bilirubin, alkaline phosphatase, uric acid, albumin, and total protein). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Number of participants with change from baseline and absolute values in QTcF meeting criteria of potential clinical concern | Baseline up to Day 12
  Federicia corrected QT (QTcF) will be summarized using actual values and changes from baseline. The participants meeting criteria of potential clinical concern will be judged by investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461040